CLINICAL TRIAL: NCT06379711
Title: Cardiopulmonary Changes Following Spinal Cord Stimulation in Individuals With Spinal Cord Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Andrei Krassioukov, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H22-03727
Record Dates: First submitted 2024-04-02; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Spinal Cord Injuries; Cardiovascular Diseases; Cardiopulmonary Diseases
Keywords: Spinal Cord Stimulation; Transcutaneous Spinal Cord Stimulation; Cardiovascular dysfunction; Cardiopulmonary dysfunction; Cardiovascular Biomarkers; Endothelial cell-derived Microvesicles; Plasma Catecholamines; Autonomic Dysreflexia; Orthostatic Hypotension
MeSH Terms: conditions — Spinal Cord Injuries; Cardiovascular Diseases; Pulmonary Heart Disease; Autonomic Dysreflexia; Hypotension, Orthostatic

STUDY DESIGN:
Intervention Model Description: Pre-Post Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcutaneous spinal cord stimulation (tSCS) (Experimental): Exploring the mechanisms of SCS for improving cardiovascular function in individuals with chronic, motor-complete SCI by measuring vascular related endothelial biomarkers and plasma catecholamines
  Interventions: Device: Transcutaneous Spinal Cord Stimulation (tSCS)

INTERVENTIONS:
Device: Transcutaneous Spinal Cord Stimulation (tSCS) — Transcutaneous spinal cord stimulation (tSCS) will be delivered via a non-invasive central nervous system stimulator TESCoN or SCONE (SpineX Inc., CA - experimental type II medical devices) through self-adhesive electrode(s) placed on the skin between spinous processes over the midline of the vertebral column as the cathode(s) and two rectangular electrodes placed symmetrically on the skin over the iliac crests as anodes. Stimulation will be applied at various waveforms and frequencies (ranging between 1Hz and 90Hz) with and without a carrier frequency. Current amplitude will start at 10mA and proceed incrementally until tolerable or responses plateau. If spasticity occurs or is uncomfortable, the current will be decreased. Specific areas for electrode placement will be examined and prepared to reduce skin impedance. tSCS will be delivered under the supervision of a physician (Dr. Krassioukov/Dr. Berger) by trained doctoral/post-doctoral trainees.
  Other Names: TESCoN device by SpineX Inc., CA, USA - experimental type II medical device; SCONE device by SpineX Inc., CA, USA - experimental type II medical device

SUMMARY:
The aim of this study is to examine the mechanisms of transcutaneous spinal cord stimulation (tSCS) for improving cardiovascular and pulmonary function in individuals with chronic motor-complete spinal cord injury (SCI) by measuring vascular related endothelial biomarkers, plasma catecholamines, and respiratory parameters.

DETAILED DESCRIPTION:
DETAILED RESEARCH PROCEDURES

(A) INFORMED CONSENT:

Prospective participants will be provided with the study informed consent form and will be given at least 24 hours to review the form, ask questions, and discuss with whomever they like.

(B) VISIT 1 -Screening

Approximately 1 hour

Individuals who agree to participate in the study will be invited for a screening assessment to confirm study eligibility. After the individual has provided informed consent, they will be assigned a unique study identification number and the information listed below will be collected.

Screening questionnaires and assessments:

* Inclusion/Exclusion Criteria confirmation
* Demographics
* Medical history and history of injury
* Concomitant medication use
* Weight and height
* Previous allergies and adverse events to medications
* Pregnancy screening will be performed
* Internationals Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) exam

(C) VISITS 2-5 -Baseline functional assessments, questionnaires, and cardiopulmonary assessments

Approximately 2 hours per visit

Enrolled participants will complete questionnaires after which a spirometry assessment for pulmonary function will be performed. Participants will be provided with a 24-hour Ambulatory Blood Pressure Monitor (24- ABPM) device to take home to record daily changes in cardiovascular parameters.

Questionnaires (Visit 2):

* Short-form (36) Health Survey (SF-36)
* Autonomic Dysfunction following SCI (ADFSCI) questionnaire
* Leisure Time Physical Activity Questionnaire after SCI (LTPAQ-SCI).
* National Health Interview Survey - Chronic Conditions
* American Thoracic Society (ATS) Adult Respiratory Disease Survey. - Tobacco Use

Baseline cardiopulmonary and optional functional assessments (with and without tSCS) (Visits 2-5):

* Spirometry testing (Visit 2)
* 24-hour Ambulatory Blood Pressure and electrocardiogram Monitoring (24-hr ABP and ECG Monitor) (Visit 2)
* Somatosensory evoked potentials (Visit 3, optional)
* Transcranial Magnetic Stimulation (Visit 4, optional)
* H-reflex (Visit 5, optional)
* Compound Muscle Action Potentials (Peripheral nerve stimulation) (Visit 5, optional)
* Muscle Ultrasound (Visit 5, optional)

Participants will also be provided with instructions to prepare for Visit 3 or 6 (depending on whether they do the optional assessments), during which blood samples will be collected. Participants will be asked to:

* Arrive for testing in a fasted state (fasted for 12 hours, but they may continue to drink water)
* Not consume caffeine, recreational drugs, alcohol, smoking, or antihypotensive drug (e.g., midodrine) for 12 hours prior to their appointment
* No strenuous exercise within 24 hours of the start of the study.

(D) VISITS 3-5 or 6-8 (depending on whether or not the optional functional assessments were completed earlier in the study). Baseline cardiovascular assessments and blood draws.

Approximately 3 hours

In this session, participants will return the 24-hour ABP and ECG Monitor and undergo baseline cardiovascular assessments as well as the blood draws. The participant has the option of only taking part in one or all cardiovascular assessments. If the participant chooses to undergo more than one cardiovascular assessment they will be conducted on different visits.

Cardiovascular Assessments:

• Cardiovascular stress test (orthostatic stress test and/or vibrostimulation or DARS)

Blood Draws:

Four (4) blood draws will be taken:

1. At rest without tSCS
2. At rest with tSCS
3. During cardiovascular stress test without tSCS
4. During cardiovascular stress test with tSCS

(E) TREATMENT VISITS (minimum 12 tSCS visits, depending on whether or not the optional functional and cardiovascular assessments were done earlier in the study) to completion of long-term intervention with tSCS intervention:

Each session will last approximately 90 minutes (set-up AND at least 45min of tSCS treatment).

Long-term tSCS is scheduled to last for a minimum of two times per week for 6 weeks.

Following the completion of the intervention, participants will begin post-intervention questionnaires and cardiopulmonary assessments. Week to week variation in the number of scheduled sessions may vary due to varying circumstances (e.g., scheduling, transportation, participant health). However, the total number of sessions conducted will be the same as the participant's original goal.

(F) SECOND TO LAST VISIT: Post-intervention questionnaires and cardiopulmonary assessment:

Approximately 2 hours

In this session, participants will complete post-intervention questionnaires and undergo post-intervention cardiopulmonary assessments.

Questionnaires:

* Short-form (36) Health Survey (SF-36)
* Autonomic Dysfunction following SCI (ADFSCI) questionnaire
* Leisure Time Physical Activity Questionnaire after SCI (LTPAQ-SCI).
* National Health Interview Survey - Chronic Conditions
* American Thoracic Society (ATS) Adult Respiratory Disease Survey. - Tobacco Use

Cardiopulmonary Assessments:

* Spirometry testing
* 24-hour ABP and ECG Monitor

(G) LAST VISIT: Post-intervention cardiovascular assessments and blood draws:

Approximately 3 hours

In this session, participants will undergo post-intervention cardiovascular assessments as well as the blood draws.

Cardiovascular Assessments:

* Carotid and cardiac ultrasound
* Cardiovascular stress test (orthostatic hypotension stress and/or vibrostimulation or DARS)

Blood Draws:

Four (4) blood draws will be taken:

1. At rest without tSCS
2. At rest with tSCS
3. During a cardiovascular stress without tSCS
4. During a cardiovascular stress with tSCS

ELIGIBILITY:
INCLUSION & EXCLUSION CRITERIA:

INCLUSION CRITERIA:

A participant must meet all of the following criteria in order to be eligible for inclusion:

1. Resident of British Columbia, Canada with active provincial medical services plan
2. Male or female, 19-65 years of age
3. Chronic SCI at or above the T10 spinal cord segment
4. >1-year post injury or diagnosis, at least 6 months from any spinal surgery.
5. American Spinal Injury Association Impairment Scale (AIS) A, B, C and D for SCI
6. Stable management of spinal cord related clinical issues (e.g., spasticity management)
7. Women of childbearing potential must not be intending to become pregnant, currently pregnant, or lactating. The following conditions apply:

   7.1 Women of childbearing potential must have a confirmed negative pregnancy test prior to the baseline visit.

   7.2 Women of childbearing potential must agree to use adequate contraception during the period of the trial and for at least 28 days after completion of treatment. Effective contraception includes abstinence.
8. Sexually active males with female partners of childbearing potential must agree to use effective contraception during the period of the trial and for at least 28 days after completion of treatment.
9. Must provide informed consent.
10. Able to understand and complete study-related questionnaires (must be able to understand and speak English or have access to an appropriate interpreter as judged by the investigator).
11. Willing and able to comply with all clinic visits and study-related procedures.

EXCLUSION CRITERIA:

A participant who meets any of the following criteria will not be eligible to participate:

1. Ventilator dependent.
2. Painful musculoskeletal dysfunction, unhealed fracture, pressure sore, or active infection that may interfere with testing
3. Clinically significant, unmanaged, depression (PHQ-9 above 15) or ongoing drug abuse.
4. Use of any medication or treatment that in the opinion of the investigator indicates that it is not in the best interest of the participant to participate in this study.
5. Intrathecal baclofen pump.
6. Cardiovascular, respiratory, bladder, or renal disease unrelated to SCI or presence of hydronephrosis or presence of obstructive renal stones.
7. Presence of severe acute medical issue(s) that in the investigator's judgement would adversely affect the participant's participation in the study (e.g., pressure sore, urinary tract infection, etc.).
8. Any implanted metal (other than dental implants) in the skull or presence of pacemakers, stimulators, or medication pumps in the trunk.
9. Severe anemia (Hgb<8 g/dl) or hypovolemia as measured by hematocrit via blood test in the last six months.
10. Participant has undergone electrode implantation surgery.
11. Participant is a member of the investigational team or his/her immediate family.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Circulating endothelial biomarkers in EMV/µL (Park et al., 2023) | Real-time Effect: 1 week; Long-term Effect: 8 weeks
  Real-time Effect: Change in circulating endothelial biomarkers (i.e., endothelial cell derived microvesicles (EMVs)) before and after real-time tSCS during cardiovascular stress (i.e., head-up tilt test to trigger orthostatic hypotension OH and/or vibrostimulation/DARS to trigger AD).
  Long-term Effect: Change from baseline in circulating endothelial biomarkers (i.e., endothelial cell derived microvesicles (EMVs)) before and after long-term tSCS intervention during cardiovascular stress (i.e., head-up tilt test to trigger OH and/or vibrostimulation/DARS to trigger AD).

SECONDARY OUTCOMES:
Plasma catecholamines in nmol/L (Claydon & Krassioukov, 2008) | Real-time Effect: 1 week; Long-term Effect: 8 weeks
  Real-time Effect: Change in plasma catecholamines (e.g., norepinephrine) before and after real-time tSCS during cardiovascular stress (i.e., head-up tilt test to trigger orthostatic hypotension OH and/or vibrostimulation/DARS to trigger AD).
  Long-term Effect: Change from baseline in plasma catecholamines (e.g., norepinephrine) before and after long-term tSCS intervention during cardiovascular stress (i.e., head-up tilt test to trigger OH and/or vibrostimulation/DARS to trigger AD).
Spirometric parameters for lung volume in ml/kg (Aung et al., 2019) for FVC | Real-time Effect: 1 week; Long-term Effect: 8 weeks
  Real-time Effect: Change in spirometric parameters (i.e., forced vital capacity (FVC)), before and after real-time tSCS during cardiovascular stress (i.e., head-up tilt test to trigger orthostatic hypotension OH and/or vibrostimulation/DARS to trigger AD).
  Long-term Effect: Change from baseline in spirometric parameters (i.e., forced vital capacity (FVC)), before and after long-term tSCS intervention during cardiovascular stress (i.e., head-up tilt test to trigger OH and/or vibrostimulation/DARS to trigger AD).
Spirometric parameters for lung volume in ml/kg (Aung et al., 2019) for FEV1 | Real-time Effect: 1 week; Long-term Effect: 8 weeks
  Real-time Effect: Change in spirometric parameters (i.e., forced expiratory volume (FEV) in 1 second (FEV1)), before and after real-time tSCS during cardiovascular stress (i.e., head-up tilt test to trigger orthostatic hypotension OH and/or vibrostimulation/DARS to trigger AD).
  Long-term Effect: Change from baseline in spirometric parameters (i.e., forced expiratory volume (FEV) in 1 second (FEV1)), before and after long-term tSCS intervention during cardiovascular stress (i.e., head-up tilt test to trigger OH and/or vibrostimulation/DARS to trigger AD).

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Krassioukov, MD,PhD,FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- Blusson Spinal Cord Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
The research team plans to deposit final de-identified research data at a community-based repository for SCI research, such as Open Data Commons for SCI (https://odc-sci.org//). Research resources, including but not limited to, established stimulation parameter and recording equipment, will also be made available through material transfer agreement upon reasonable request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available upon full-text print publication in a peer-reviewed journal, for a duration of at least 10 years.
Access Criteria: Online access or e-mail request to the corresponding author from an established scientific investigator.

REFERENCES:
- [Background] Hubli M, Gee CM, Krassioukov AV. Refined assessment of blood pressure instability after spinal cord injury. Am J Hypertens. 2015 Feb;28(2):173-81. doi: 10.1093/ajh/hpu122. Epub 2014 Jul 1. PMID 24990527
- [Background] Forchheimer M, McAweeney M, Tate DG. Use of the SF-36 among persons with spinal cord injury. Am J Phys Med Rehabil. 2004 May;83(5):390-5. doi: 10.1097/01.phm.0000124441.78275.c9. PMID 15100631
- [Background] The National Health Interview Survey design, 1973-84, and procedures, 1975-83. Vital Health Stat 1. 1985 Aug;(18):1-127. No abstract available. PMID 4082502
- [Background] Ferris BG. Epidemiology Standardization Project (American Thoracic Society). Am Rev Respir Dis. 1978 Dec;118(6 Pt 2):1-120. No abstract available. PMID 742764
- [Background] Martin Ginis KA, Phang SH, Latimer AE, Arbour-Nicitopoulos KP. Reliability and validity tests of the leisure time physical activity questionnaire for people with spinal cord injury. Arch Phys Med Rehabil. 2012 Apr;93(4):677-82. doi: 10.1016/j.apmr.2011.11.005. Epub 2012 Feb 13. PMID 22336103
- [Background] Consortium for Spinal Cord Medicine. Early acute management in adults with spinal cord injury: a clinical practice guideline for health-care professionals. J Spinal Cord Med. 2008;31(4):403-79. doi: 10.1043/1079-0268-31.4.408. No abstract available. PMID 18959359
- [Background] Hubli M, Krassioukov AV. Ambulatory blood pressure monitoring in spinal cord injury: clinical practicability. J Neurotrauma. 2014 May 1;31(9):789-97. doi: 10.1089/neu.2013.3148. Epub 2014 Jan 30. PMID 24175653
- [Background] Standardization of Spirometry, 1994 Update. American Thoracic Society. Am J Respir Crit Care Med. 1995 Sep;152(3):1107-36. doi: 10.1164/ajrccm.152.3.7663792. No abstract available.
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Pithon KR, Martins LE, Renno AC, Abreu DC, Cliquet A Jr. Pulmonary function testing in quadriplegic subjects. Spinal Cord. 2008 Apr;46(4):275-7. doi: 10.1038/sj.sc.3102146. Epub 2007 Nov 20. PMID 18026172
- [Background] Kelley A, Garshick E, Gross ER, Lieberman SL, Tun CG, Brown R. Spirometry testing standards in spinal cord injury. Chest. 2003 Mar;123(3):725-30. doi: 10.1378/chest.123.3.725. PMID 12628869
- [Background] Park AJ, Fandl HK, Garcia VP, Coombs GB, DeSouza NM, Greiner JJ, Barak OF, Mijacika T, Dujic Z, Ainslie PN, DeSouza CA. Differential Expression of Vascular-Related MicroRNA in Circulating Endothelial Microvesicles in Adults With Spinal Cord Injury: A Pilot Study. Top Spinal Cord Inj Rehabil. 2023 Spring;29(2):34-42. doi: 10.46292/sci22-00032. Epub 2023 Apr 3. PMID 37235195
- [Background] Claydon VE, Krassioukov AV. Clinical correlates of frequency analyses of cardiovascular control after spinal cord injury. Am J Physiol Heart Circ Physiol. 2008 Feb;294(2):H668-78. doi: 10.1152/ajpheart.00869.2007. Epub 2007 Nov 16. PMID 18024546
- [Background] Aung HH, Sivakumar A, Gholami SK, Venkatewaran SP, Gorain B, Shadab M. An overview of the anatomy and physiology of the lung, in Nanotechnology-Based Targeted Drug Delivery Systems for Lung Cancer, 2019; 1-20.